CLINICAL TRIAL: NCT05682404
Title: Prevalence, Associated Factors Points and Implementation of Care Procedures of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation in Healthcare Institution. Prospective Cohort Study
Brief Title: Prevalence, Associated Factors Points and Implementation of Care Procedures of Chronic Obstructive Pulmonary Disease Exacerbation in Healthcare Institution
Acronym: OPEDEXA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: OPEDEXA (38RC17.073)
Record Dates: First submitted 2019-04-16; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: COPD Exacerbation
Keywords: COPD; exacerbation; Prospective; Observational; Professional practices guidelines
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a public health problem responsible for high mortality rate and significant costs for society. The disease evolution is punctuated by exacerbations worsening the health state of patients.

Many guidelines of care procedures have been written but many disparities persist in medical practices.

This pilot prospective observational study is an overview of current local practices in the university health center of Grenoble Alpes and it is the first step towards developing a regional observatory in order to standardize and improve patient cares. The primary outcome is to compare the international guidelines to the local practices regarding the prescription of key treatments of exacerbation, especially antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years (included)
* Known or suspected Chronic Obstructive Pulmonary Disease
* Admitted for COPD exacerbation in emergency department or pneumology department or intensive care unit of university health center of Grenoble Alpes during the period of data collection.

Exclusion Criteria:

* opposition to participate at the study
* Patients under the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every Patient who is admitted for COPD exacerbation in emergency department or pneumology department or intensive care unit of university health center of Grenoble Alpes during the period of data collection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of antibiotics prescriptions following the guidelines in COPD exacerbation. | up to 30 days
  Adherence to guidelines regarding antibiotics prescription in COPD exacerbation that is justified by :
  * sputum purulence
  * severe symptoms
  * severe comorbidities
  * pneumonia

SECONDARY OUTCOMES:
Percentage of corticosteroids prescriptions following the guidelines in COPD exacerbation. | up to 30 days
  Adherence to guidelines regarding corticosteroids prescription in COPD exacerbation that is :
  * not a systematic prescription
  * if needed, it is 30 to 40mg per day of prednisone equivalent and 5 to 7 days maximum
Percentage of hospitalization of patients following the guidelines in COPD exacerbation. | up to 30 days
  Adherence to guidelines regarding hospitalization criteria in COPD exacerbation that are :
  * severe symptoms
  * respiratory failure
  * failure of first treatments
  * severe comorbidities
  * deficient social environment
  * patient older than 85 years old
  * baseline dyspnea around 4 to 5 in Modified Medical Research Council Dyspnea Scale (mMRC scale)
  Adherence to guidelines regarding criteria for intensive care unit hospitalization in COPD exacerbation that are :
  * severe dyspnea not responding to first treatments
  * neurologic troubles
  * persistant hypoxemia despite oxygen administration or Non Invasive Ventilation.
  * respiratory acidosis despite Non Invasive Ventilation
  * need for invasive mechanical ventilation
  * hemodynamic instability and need for aminergic support
Percentage of non invasive ventilation following the guidelines in COPD exacerbation. | up to 30 days
  Adherence to guidelines regarding criteria for non invasive ventilation in COPD exacerbation that are :
  * respiratory acidosis
  * signs of respiratory failure
  * hypoxemia despite oxygen administration
  * absence of medical contraindications
Percentage of invasive ventilation following the guidelines in COPD | up to 30 days
  Adherence to guidelines regarding criteria for invasive ventilation in COPD exacerbation that are :
  * failure of non invasive ventilation
  * medical contraindications for non invasive ventilation
  * cardiac arrest
  * neurologic troubles needing sedation
  * pernicious vomiting
  * ineffective coughing
Percentage of minimal medical examinations following the guidelines in COPD exacerbation. | up to 30 days
  Adherence to guidelines regarding the prescription of minimal medical examinations in COPD exacerbation that is :
  * complete blood count, kidney function, glucose level
  * blood gases
  * chest radiography
  * electrocardiogram
  * bacteriological sputum examination only if antibiotic-resistant germ infection is suspected.
Percentage of follow-up management after COPD exacerbation following the guidelines | up to 30 days
  Adherence to guidelines regarding follow-up management after COPD exacerbation that is :
  * adherence to discharge criteria
  * first medical evaluation one week after discharge
  * early specialized follow-up into four to six weeks after discharge
Frequency of advance directives. | at day 0
  Frequency of advance directives written by patients with COPD

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France